CLINICAL TRIAL: NCT05883839
Title: Turkish Validity and Reliability Study of the "Sexual Health Care Questionnaire" for Nursing Students
Brief Title: Turkish Validity and Reliability Study of the "Sexual Health Care Questionnaire"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, CEYDA SU GUNDUZ, Study director, Marmara University
Other Study IDs: marmaraceydasugunduzistanbul
Record Dates: First submitted 2023-04-07; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Nursing Education; Nursing Students; Sexuality; Sexual Health; Validation Study
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Student Group: Three scales (knowledge, attitude, self-efficacy) in the "Sexual Healthcare Questionnaire" will be applied to 2nd and 3rd year nursing students. The scales will be re-administered to at least 30 students within 4 weeks.
  Interventions: Other: Student Group

INTERVENTIONS:
Other: Student Group — "Sexual Healthcare Questionnaire" will be applied to nursing students to adapt it to Turkish.

SUMMARY:
Determining the knowledge, attitudes and self-efficacy of nursing students in the field of sexual health care is important for the development and planning of nursing education and research. There is no Turkish tool in the literature that will enable a comprehensive assessment of nursing students' knowledge, attitudes and self-efficacy towards sexual health care. The aim of the study is to determine the validity and reliability of the Turkish version of the three scales (knowledge, attitude, self-efficacy) in the "Sexual Healthcare Questionnaire" for nursing students. This is a methodological study. These scales translated into Turkish language. Data will be collected in April 2023 through an online questionnaire from nursing students at a public university in Turkey. The test-retest will be performed again after 4 weeks. At least 310 participants from 2nd and 3rd year nursing students will be included in the study.

DETAILED DESCRIPTION:
Sexuality is an indispensable part of being human, affecting the lives of individuals. It is necessary to provide sexual health services to support the quality of life of individuals who have problems with sexual health. In addition to being in a unique position in the field of practice to provide sexual health care, nurses' service on sexual issues is an important professional responsibility in order to provide holistic care. Determining the knowledge, attitudes and self-efficacy of nursing students in the field of sexual health care is important for the development and planning of nursing education and research. There is no Turkish tool in the literature that will enable a comprehensive assessment of nursing students' knowledge, attitudes and self-efficacy towards sexual health care. The aim of the study is to determine the validity and reliability of the Turkish version of the three scales (knowledge, attitude, self-efficacy) in the "Sexual Healthcare Questionnaire" for nursing students. This is a methodological study. These scales translated into Turkish language. Data will be collected in April 2023 through an online questionnaire from nursing students at a public university in Turkey. The test-retest will be performed again after 4 weeks. At least 310 participants from 2nd and 3rd year nursing students will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd or 3rd year nursing student
* Absence of psychiatric illness
* Being willing to participate

Exclusion Criteria:

* Desire to leave the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 310 students should form the sample size, which is 10 times the "Knowledge of Sexual Healthcare Scale", which has the highest number of items with 31 items among the scales in our survey.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Sexual Healthcare Scale | baseline
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Knowledge of Sexual Healthcare Scale | Retest (later 4 weeks)
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Attitude to Sexual Healthcare Scale | baseline
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 sub-dimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.
Attitude to Sexual Healthcare Scale | Retest (later 4 weeks)
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 sub-dimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.
Self-Efficacy for Sexual Healthcare Scale | baseline
  The scale measures nursing students' self-efficacy in providing sexual health services. The scale consists of 3 sub-dimensions and a total of 22 items. Each item is rated on a 5-point Likert scale ranging from 1= strongly disagree, 2= disagree, 3= undecided, 4= agree, 5= strongly agree. The total score ranges from 22 to 110 points.
Self-Efficacy for Sexual Healthcare Scale | Retest (later 4 weeks)
  The scale measures nursing students' self-efficacy in providing sexual health services. The scale consists of 3 sub-dimensions and a total of 22 items. Each item is rated on a 5-point Likert scale ranging from 1= strongly disagree, 2= disagree, 3= undecided, 4= agree, 5= strongly agree. The total score ranges from 22 to 110 points.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Demirci, Prof., Study Director — Marmara Üniversity
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No